CLINICAL TRIAL: NCT04938232
Title: A Phase II Trial of Ipilimumab With and Without Nivolumab in Patients With Relapsed/Refractory Classic Hodgkin Lymphoma
Brief Title: Ipilimumab With or Without Nivolumab in Relapsed/Refractory cHL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Reid Merryman, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-204
Record Dates: First submitted 2021-06-08; First posted 2021-06-24 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Hodgkin Lymphoma; Relapsed Hodgkin's Disease, Adult; Refractory Hodgkin Lymphoma
Keywords: Hodgkin lymphoma; Relapsed Hodgkin's Disease, Adult; Refractory Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Disease Progression after previous therapy (Experimental): Participants will receive Ipilimumab alone and depending on response will receive either a maintenance course of Ipilimumab or a course of Nivolumab and Ipilimumab in combination followed by a maintenance course of Ipilimumab. Patients who have progressive disease after fewer than 4 cycles of ipilimumab are also eligible to proceed to combination therapy with nivolumab and ipilimumab, if they are clinically stable.
  * Ipilimumab Monotherapy: Every 3 weeks for 4 study cycles
  * Complete Response/Partial Response: Maintenance Ipilimumab every 12 weeks for 8 cycles
  * Stable or Progressive Disease Response: Nivolumab and Ipilimumab every 3 weeks for 4 study cycles, followed by Maintenance Ipilimumab every 12 weeks for 7 cycles
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Intravenous infusion
  Other Names: Opdivo
Drug: Ipilimumab — Intravenous infusion
  Other Names: Yervoy

SUMMARY:
This study is looking at the effects of Ipilimumab when it is given alone or in combination with Nivolumab to patients with relapsed or refractory classic Hodgkin's lymphoma (cHL).

The names of the study drugs involved in this study are:

* Ipilimumab
* Nivolumab

DETAILED DESCRIPTION:
This is an open-label, multi-center, phase II study of ipilimumab with or without nivolumab for patients with relapsed or refractory (R/R) classic Hodgkin lymphoma (cHL).

Nivolumab is a drug which is approved by the United States Food and Drug Administration (FDA) for the treatment of adult patients experiencing relapsed Hodgkin lymphoma (cHL) who have received at least two prior systemic therapies.

Ipilimumab has been approved by the FDA for the treatment of metastatic melanoma (a type of skin cancer), and specific types of previously treated advanced kidney cancers.

The study drugs have not been approved in combination for cHL by the Food and Drug Administration (FDA). This study is for participants who previously had progressive disease when receiving a PD-1 mAb.

Participants will receive 4 cycles of ipilimumab monotherapy and then undergo restaging imaging. Patients who achieved an objective response will continue treatment with ipilimumab maintenance. Other patients will receive 4 cycles of nivolumab and ipilimumab followed by ipilimumab maintenance treatment. Patients who have progressive disease after fewer than 4 cycles of ipilimumab are eligible to proceed to combination therapy with nivolumab and ipilimumab if they are clinically stable. Participants will receive up to ~ 24 months of study treatment.

After completion of therapy, participants will be followed every 3 months for 2 years and then every 6 months for the next 5 years.

It is expected that about 13 people will participate in this research study.

Bristol Myers Squibb (BMS) is supporting this research study by providing the study drugs and funding for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically determined classic Hodgkin lymphoma with pathologic review at the participating institution.
* Participants must have measurable disease, defined as a lymph node or tumor mass ≥1.5 cm in at least one dimension by CT, PET/CT, or MR. Imaging must have been completed no greater than 6 weeks prior to study enrollment. Measurable disease that has previously been irradiated is permissible only if there has been evidence of progression since the radiation.
* Patients must have progressed after two or more lines of systemic treatment, including autologous stem cell transplantation, if eligible.
* Progression of disease or relapse following treatment with nivolumab or pembrolizumab. Intervening treatments with between PD-1 mAb therapy and the trial are permitted.
* Patients may have had a prior autologous stem cell transplant and may have been treated with chimeric antigen receptor T-cells (CAR T-cells).
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (see Appendix A)
* Adequate hematologic and organ function as defined below:

  * Absolute neutrophil count > 1.0x109/L unless due to marrow involvement by lymphoma in which case ANC must be >0.75x109/L. Growth factor support is allowed provided it is received at least 5 days prior to enrollment labs.
  * Platelets > 75 x109/L, unless due to marrow involvement by lymphoma, in which case platelets must be >50 x109/L
  * Estimated GFR (by Cockroft-Gault equation) > 40ml/min
  * Total bilirubin < 1.5 X ULN
  * AST/ALT < 2.5 X ULN
* Ability to understand and the willingness to sign a written informed consent document.
* Willingness to provide pre-treatment tumor sample by core needle or excisional surgical biopsy. An archival sample is acceptable in the following situations: the sample was acquired within 90 days of initiation of PD-1 therapy AND the following provisions are met: 1) availability of a tumor-containing formalin fixed, paraffin embedded (FFPE) tissue block, 2) if the tumor containing FFPE tissue block cannot be provided in total, sections from this block should be provided that are freshly cut and mounted on positively charged glass slides (SuperFrost Plus are recommended). Preferably, 25 slides should be provided; if not possible, a minimum of 15 slides is required. Exceptions to this criterion may be made with approval of the Study Chair.
* Willingness to use contraception during and after study treatment. Women of child-baring potential (WOCBP) will be instructed to adhere to contraception for a period of 5 months following last dose of nivolumab and 6 months following the last dose of ipilimumab. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after last dose of nivolumab and 6 months after the last dose of ipilimumab.

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 28 days of the start of study drug (including chemotherapy, radiation therapy, antibody-based therapy, etc.), or 56 days for radioimmunotherapy. Steroids for symptom palliation are allowed but must be either discontinued or on stable doses of < 10mg daily of prednisone (or the equivalent) at the time of initiation of protocol therapy.
* Patients may not be receiving any other investigational agents or have received investigational agents within 4 weeks (or 3 half-lives, whichever is longer) of beginning treatment.
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy unless in consultation with an allergy specialist they are deemed eligible for retreatment with desensitization.
* Patients who have undergone prior allogeneic stem cell transplantation
* Patients with a history of or active autoimmune disease (except controlled asthma, Hashimoto thyroiditis, atopic dermatitis, or vitiligo), or requiring systemic corticosteroids at a dose of 10mg prednisone equivalent daily. Patients with a history of autoimmune disease who never required corticosteroids and with no evidence of disease activity, and in whom the risk of reactivation is felt not to be serious, may be enrolled after discussion with the overall study chair. Exceptions to this are patients with a history of inflammatory bowel disease (ulcerative colitis and Crohn's disease). These patients are excluded regardless of whether their disease is active or inactive.
* Patients who experienced grade 4 immune-related adverse events (irAEs) during treatment with a PD-1 mAb.
* Patients with active pneumonitis or colitis, or patients with cirrhosis.
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia).
* Patients with known HIV infection or hepatitis B or C infection. Testing for HIV is optional. Testing for hepatitis B and C is mandatory. Patients with hepatitis B core Ab positivity but negative surface antigen and negative viral load may be enrolled if they can be treated with a prophylactic agent (eg, entecavir); patients with hepatitis C seropositivity who have a negative viral load can also be enrolled.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Prior history of another malignancy (except for non-melanoma skin cancer or in situ cervical or breast cancer) unless disease free for at least 2 years. Patients with prostate cancer are allowed if PSA is less than 1.
* Patients should not have received immunization with attenuated live vaccine within one week of study entry or during study period.
* History of noncompliance to medical regimens.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study.
* Patients with any one of the following currently on or in the previous 6 months will be excluded: myocardial infarction, congenital long QT syndrome, torsade de pointes, left anterior hemiblock, unstable angina, coronary/peripheral artery bypass graft, or cerebrovascular accident.
* Other uncontrolled intercurrent illness that would limit adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2026-08-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Reid W Merryman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - University of Chicago Medicine, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Disease Progression After Previous Therapy: Participants will receive Ipilimumab alone and depending on response will receive either a maintenance course of Ipilimumab or a course of Nivolumab and Ipilimumab in combination followed by a maintenance course of Ipilimumab. Patients who have progressive disease after fewer than 4 cycles of ipilimumab are also eligible to proceed to combination therapy with nivolumab and ipilimumab, if they are clinically stable.
  * Ipilimumab Monotherapy: Every 3 weeks for 4 study cycles
  * Complete Response/Partial Response: Maintenance Ipilimumab every 12 weeks for 8 cycles
  * Stable or Progressive Disease Response: Nivolumab and Ipilimumab every 3 weeks for 4 study cycles, followed by Maintenance Ipilimumab every 12 weeks for 7 cycles
  Nivolumab: Intravenous infusion
  Ipilimumab: Intravenous infusion
Period: Overall Study
Arm/Group | Disease Progression After Previous Therapy
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 39 [23 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13
ECOG Performance Status Scale [Count of Participants; unit: Participants]
  0 - Fully active | 6
  1 - Restricted in physically strenuous activity | 6
  2 - Ambulatory and capable of all selfcare but unable to carry out any work activities | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Patients achieving a complete (CR) or partial response (PR), assessed by PET/CT (using Lugano)
Time Frame: From enrollment to completion of 4 cycles (each cycle is 21 days) of treatment
Measure: Number (90% Confidence Interval); unit: percent
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 13
percent | 23 [7 to 49]

2. Secondary Outcome: Overall Response Rate (ORR) Ipilimumab Monotherapy, Lugano
Description: Patients achieving complete (CR) or partial response (PR), assessed by PET/CT (using Lugano criteria) after ipilimumab monotherapy
Time Frame: 12 weeks
Measure: Number (90% Confidence Interval); unit: percent
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 13
percent | 23 [7 to 49]

3. Secondary Outcome: Overall Response Rate (ORR) Ipilimumab Monotherapy, LYRIC
Description: Patients achieving complete (CR) or partial response (PR), assessed by PET/CT (using LYRIC criteria) after ipilimumab monotherapy
Time Frame: 12 weeks
Measure: Number (90% Confidence Interval); unit: percent
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 13
percent | 23 [7 to 49]

4. Secondary Outcome: Complete Response Rate (CRR) Ipilimumab Monotherapy, Lugano
Description: Patients achieving complete response (CR), assessed by PET/CT (using Lugano criteria) after ipilimumab monotherapy
Time Frame: 12 weeks
Measure: Number (90% Confidence Interval); unit: percent
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 13
percent | 0 [0 to 21]

5. Secondary Outcome: Complete Response Rate (CRR) Ipilimumab Monotherapy, LYRIC
Description: Patients achieving complete response (CR), assessed by PET/CT (using Lugano criteria) after ipilimumab monotherapy
Time Frame: 12 weeks
Measure: Number (90% Confidence Interval); unit: percent
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 13
percent | 0 [0 to 21]

6. Secondary Outcome: Overall Response Rate (ORR) Ipilimumab and Nivolumab Combination Therapy, Lugano
Description: Patients achieving complete (CR) or partial response (PR), assessed by PET/CT (using Lugano criteria) after ipilimumab and nivolumab combination therapy
Time Frame: 24 weeks
Measure: Number (90% Confidence Interval); unit: percent
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 13
percent | 15 [3 to 41]

7. Secondary Outcome: Overall Response Rate (ORR) Ipilimumab and Nivolumab Combination Therapy, LYRIC
Description: as for outcome 6
Time Frame: 24 weeks
Measure: Number (90% Confidence Interval); unit: percent
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 13
percent | 8 [0 to 32]

8. Secondary Outcome: Progression-free Survival, LYRIC
Description: Percent of patients alive and progression-free at 2-years. Time from registration to progression or death, censored at date last known alive and progression-free using LYRIC criteria
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 13
percent | 38 [14 to 97]

9. Secondary Outcome: Duration of Response
Description: 2-year percent DOR using Lugano criteria (LYRIC was equivalent). Time from first response (PR or CR) to progression, censored at last disease assessment.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 3
percent | 100 [100 to 100]

10. Secondary Outcome: Progression-free Survival, Lugano
Description: Percent of patients alive and progression-free at 2-years. Time from registration to progression or death, censored at date last known alive and progression-free using Lugano criteria
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 13
percent | 49 [24 to 99]

11. Secondary Outcome: Overall Survival
Description: Percent OS at 2-years. Time from registration to death from any cause, censored at date last known alive
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 13
percent | 75 [43 to 100]

12. Secondary Outcome: Percent of Patients With Grade 3+ Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0
Description: Worst grade adverse event attributable (possibly, probably, definitely) to study treatment. Descriptions and grading scales per NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Time Frame: 2 years
Measure: Number (90% Confidence Interval); unit: percent
Arm/Group | Disease Progression After Previous Therapy
Number analyzed (Participants) | 13
percent | 46 [22 to 71]

ADVERSE EVENTS:
Time Frame: 120 weeks
Arm/Group | Disease Progression After Previous Therapy
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disease Progression After Previous Therapy (N=13)
Alanine aminotransferase increased (Investigations) | 1 (3)
Lung infection (Infections and infestations) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disease Progression After Previous Therapy (N=13)
Fever (General disorders) | 8 (11)
Anemia (Blood and lymphatic system disorders) | 5 (10)
Fatigue (General disorders) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Alanine aminotransferase increased (Investigations) | 6 (6)
Alkaline phosphatase increased (Investigations) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 4 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Dizziness (Nervous system disorders) | 3 (4)
Flu like symptoms (General disorders) | 2 (4)
Headache (Nervous system disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (4)
Platelet count decreased (Investigations) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Chills (General disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3)
Hypothyroidism (Endocrine disorders) | 2 (3)
Infections and infestations - Other, specify (Infections and infestations) | 2 (3) — Bilateral hand rash (n=1), Covid-19 infection (n=1), strep throat (n=1)
Lipase increased (Investigations) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (3) — diffuse red rash (n=1), left neck biopsy site (n=1), psoriasis (n=1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Bloating (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Weight loss (Investigations) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
CPK increased (Investigations) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) — Nocturia (n=1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonia (n=1)
Shingles (Infections and infestations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Thyroid stimulating hormone increased (Investigations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT04938232/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT04938232/ICF_001.pdf